CLINICAL TRIAL: NCT06224829
Title: Characterizing Responses to Massage in Individuals With Neck Pain
Brief Title: Response to Massage in Neck Pain
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Florida (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRB202301891
Record Dates: First submitted 2024-01-16; First posted 2024-01-25 (Actual); Last update posted 2025-07-24 (Actual); Status verified 2025-07

CONDITIONS: Neck Pain
MeSH Terms: conditions — Neck Pain

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Pain Inducing Massage (Experimental): Participants will receive 60 seconds of manual pressure applied to one point in their neck followed by 30 seconds of complete pressure release 4 times for a total contact time of 240 seconds. Pressure will be applied such that the participant rates the pain = 5/10 on an 11-point numeric pain rating scale with 0 indicating no pain and 10 indicating the most severe pain imaginable.
  Interventions: Procedure: Pain Inducing Massage
- Pain Free Massage (Active Comparator): Participants will receive 60 seconds of manual pressure applied to one point in their neck followed by 30 seconds of complete pressure release 4 times for a total contact time of 240 seconds. Pressure will be applied such that the participant rates the pain = 0/10 on an 11-point numeric pain rating scale with 0 indicating no pain and 10 indicating the most severe pain imaginable.
  Interventions: Procedure: Pain Free Massage
- Cold Water Bath (Active Comparator): Participants will place their non-dominant hand into water cooled by a refrigeration unit (NESLAB RTE 7 Digital One, Thermo Scientific Co., Massachusetts, USA) that circulates water continuously to maintain a constant temperature of 6 degrees Celsius (males) or 8 degrees Celsius (females). The participant will place his or her hand in the cooled water for 60 seconds followed by a 30 second break in which the participant will remove his or her hand from the water. This will occur 4 times for a total immersion time of 240 seconds.
  Interventions: Procedure: Cold Water Bath

INTERVENTIONS:
Procedure: Pain Inducing Massage — 60 seconds of direct pressure to the neck resulting in 5/10 pain . This will be repeated four times for a total of 240 seconds
  Arms: Pain Inducing Massage
Procedure: Pain Free Massage — 60 seconds of direct pressure to the neck resulting in 0/10 pain . This will be repeated four times for a total of 240 seconds
  Arms: Pain Free Massage
Procedure: Cold Water Bath — Participants will place their hand in a cold water bath maintained at 6 to 8 degrees Celsius for 60 seconds. This will be repeated four times for a total of 240 seconds.
  Arms: Cold Water Bath

SUMMARY:
This study is interested in whether baseline measures of pain sensitivity i.e. the amount of pressure required to feel pain predicts pain relief following a pain inducing massage AND whether pain relief following a pain inducing massage is different than a pain free massage or placing your hand in a cold water bath. Participants with neck pain will be randomly assigned to receive a pain inducing massage, pain free massage, or to place their hand in a cold water bath.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 to 60 years old
* Currently experiencing neck pain with or without arm pain
* Neck pain symptom intensity rated as 4/10 or higher during the last 24 hours
* Neck pain for greater than or equal to 3 months

Exclusion Criteria:

* Non- English speaking
* Systemic medical conditions known to affect sensation (e.g. diabetes)
* History of neck surgery or fracture within the past 6 months
* Current history of chronic pain condition other than neck pain
* Diagnosis of cervical radiculopathy or cervical myelopathy
* History of whiplash
* Currently using blood thinning medication
* Any blood clotting disorder such as hemophilia
* Any contraindication to application of ice, such as: uncontrolled hypertension, cold urticaria, cryoglobulinemia, paroxysmal cold hemoglobinuria, and circulatory compromise
* Pregnancy

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 53 (Estimated)
Dates: Start 2024-04-08 (Actual); Primary Completion 2026-07-22 (Estimated); Study Completion 2026-07-22 (Estimated)

PRIMARY OUTCOMES:
Pressure Pain Threshold | Baseline and immediately following the intervention
  Pressure applied to the web space of the foot with a digital pressure algometer applied at 1 kg/s. Participants will be instructed to indicate when the sensation first changes from pressure to pain (pain threshold)

SECONDARY OUTCOMES:
Numeric Pain Rating Scale Resting Pain | Baseline, immediately following intervention
  Participants will rate their "current" neck pain on a 0 to 100 scale with 0= no pain and 100= the most intense pain imaginable
Numeric Pain Rating Scale Movement Evoked Pain | Baseline, immediately following intervention
  Participants will rate their neck pain on a 0 to 100 scale with 0= no pain and 100= the most intense pain imaginable during active cervical spine range of motion. The average rating across all motions (flexion, extension, left and right sidebend, left and right rotation) will be used in the analysis.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Florida, Gainesville, Florida, United States